CLINICAL TRIAL: NCT06749990
Title: Risk and Protective Factors for Relapse to Alcohol Use in Patients With Alcohol-related Liver Disease and Undergoing Orthotopic Liver Transplantation
Brief Title: Risk and Protective Factors for Relapse to Alcohol Use in Patients With Liver Disease Undergoing Liver Transplantation
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RICADUTA
Record Dates: First submitted 2024-11-28; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Related Liver Disease; Orthotopic Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, monocentric study, consisting of both a retrospective and a prospective component. The aim of the study is to identify risk and protective factors for alcohol relapse in patients with alcohol-related liver disease (ARLD) who have undergone orthotopic liver transplantation (OLT).

DETAILED DESCRIPTION:
For the retrospective part of the study, clinical data will be collected and analyzed from patients diagnosed with ARLD and with components of exotoxicity who underwent liver transplantation in the past five years. This data will be obtained from patient medical records, including results from laboratory tests and multidisciplinary outpatient consultations conducted as part of routine clinical practice.

The prospective phase of the study will involve the consecutive enrollment of patients diagnosed with ARLD or with exotoxicity-related etiological components who are undergoing liver transplantation at the IRCCS AOUBO. Four patient assessment points are planned, which will take place during routine follow-up visits already scheduled as part of the patient's care pathway. During these visits, data will be collected on the patient's medical history, laboratory and/or histological results, as well as diagnostic and surgical information. Additionally, through the administration of clinical questionnaires, data will be gathered on the patient's psychiatric-psychological status, history of exotoxicity, and psychosocial background.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent
* Candidates for liver transplantation due to liver disease with alcohol-related etiology (either mono- or multifactorial)
* For the retrospective part: patients who underwent OLT for ARLD during the time frame 2017-2022

Exclusion Criteria:

* Major psychopathologies and active psychoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in the retrospective cohort include those diagnosed with ARLD and exotoxicity-related components who underwent liver transplantation and were followed at the Internal Medicine Department for the treatment of severe organ failure at IRCCS AOUBO between 01/01/2017 and 31/12/2022.
  The patients in the prospective cohort are those diagnosed with ARLD or with exotoxicity-related etiologies who are referred to the Internal Medicine Department for the treatment of severe organ failure.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
alcohol relapse rate | 7 years
  To describe the population undergoing liver transplantation with a diagnosis of ARLD and exotoxicity-related components in terms of alcohol relapse rate
alcohol recurrence rate | 7 years
  To describe the population undergoing liver transplantation with a diagnosis of ARLD and exotoxicity-related components in terms of alcohol recurrence rate
Clinical data to assess the risk of alcohol relapse | 7 years
  Collection of clinical data on liver disease through routine visits to assess the risk of alcohol relapse at 12 months post-OLT
psychiatric evaluation to assess the risk of alcohol relapse | 7 years
  Administration of a clinimetric assessment composed of psychometric, self-assessment tests, already validated and widely used in the literature

SECONDARY OUTCOMES:
Impact of alcohol relapse/recurrence on liver transplant outcomes | 7 years
  To assess the impact of alcohol relapse/recurrence on liver transplant outcomes.
Identifying Risk and Protective Factors for Alcohol Relapse | 7 years
  To identify potential risk and protective factors for alcohol relapse and, consequently, to develop a multiparametric/multimodal operational model for evaluating candidates for liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Morelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy